CLINICAL TRIAL: NCT06715657
Title: Effect of Propofol Administration Time on the Incidence and Severity of Intrathecal Morphine-induced Pruritus in Parturient Undergoing Elective Cesarean Delivaries: A Prospective, Randomized, Comparative Controlled Study
Brief Title: Effect of Propofol Administration Time on the Incidence and Severity of Intrathecal Morphine-induced Pruritus in Parturient Undergoing Elective Cesarean Delivaries
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Essam Elsayed Mohamed, resident doctor at Anaesthesia ,Intensive care & pain management Faculty of Medicine, Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: propofol pruritus incidence CS
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Cesarean Section
Keywords: propofol administration time; intrathecal morphine-induced pruritus
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group A (Experimental): Patients will receive 0.5 mg/kg propofol diluted in 10 ml saline 0.9% IV injection 15 min before the end of surgery
  Interventions: Drug: Morphine intrathecal; Drug: propofol
- Group B (Experimental): Patients will receive 0.5 mg/kg propofol diluted in 10 ml saline 0.9% IV injection just before intrathecal anaesthesia
  Interventions: Drug: Morphine intrathecal; Drug: propofol
- Group C (Placebo Comparator): patients will receive intrathecal anaesthesia with morphine without other intervention
  Interventions: Drug: Morphine intrathecal

INTERVENTIONS:
Drug: Morphine intrathecal — patients intrathecal anaesthesia with morphine
Drug: propofol — patients will receive 0.5 mg/kg propofol diluted in 10 ml saline 0.9% IV injection 15 min before the end of surgery
  Arms: Group A
Drug: propofol — patients will receive 0.5 mg/kg propofol diluted in 10 ml saline 0.9% IV injection just before intrathecal anaesthesia
  Arms: Group B

SUMMARY:
Our hypothesis suggests that Administration time of intravenous propofol may affect Pruritus incidence and severity that occur after intrathecal morphine in parturient undergoing elective cesarean section (CS). the aim of the study is to investigate effect of prophylactic administration of intravenous sub-hypnotic dose of propofol before intrathecal morphine compared with the administration after intrathecal morphine on intrathecal morphine-induced pruritus incidence and severity in parturient undergoing elective cesarean delivaries.

DETAILED DESCRIPTION:
Neuraxial Anaesthesia is a frequent anaesthetic approach for cesarean delivery and other lower abdominal and lower limb anaesthetic procedures. Neuraxial morphine addition to local anaesthetic provides an effective and prolonged postoperative analgesia, but has been associated with a frequent incidence of pruritus and postoperative nausea and vomiting (PONV).

Neuraxial opioids are thought to act on central nervous system pathways to cause pruritus. Although precise mechanisms are incompletely understood, Numerous interventions have been investigated to prevent opioid-induced pruritus in the peripartum period as: Opioid receptor agonist-antagonists, Serotonin receptor antagonists.

There is dense concentration of opioid receptors and 5-HT3 receptors in the dorsal part of the spinal cord and nucleus of the spinal tract of the trigeminal nerve in the medulla. Activation of these receptors by neuraxial opioid administration or by circulating estrogen in parturient results in pruritus which is usually localized to face, neck, or upper thorax.

Propofol exerts its antipruritic action through inhibition of the posterior horn transmission in spinal cord. Series of clinical trials have reported that a sub-hypnotic dose of propofol is equally effective in reducing the incidence of pruritus following intrathecal morphine. however these studies have limited information about dose and timing of administration of propofol.

ELIGIBILITY:
Inclusion Criteria:

* Parturient of American Society of Anaesthesiologists (ASA) class I or II physical status.
* Age: 20-40 years.
* At term gestation (≥ 37 weeks) with a singleton uncomplicated pregnancy.
* Elective cesarean delivery under intrathecal anaesthesia

Exclusion Criteria:

* Parturient refusal.

  * Significant organ dysfunctions (e.g., cardiac, respiratory, renal, or liver disorders).
  * Morbid obesity (BMI >35).
  * Parturient with known hypersensitivity to propofol, morphine or amide local anaesthetics.
  * Parturient with pruritogenic systemic disease.
  * A coexisting skin disorder or preexisting pregnancy induced pruritus.
  * Parturient with any contraindication for intrathecal anaesthesia, e.g. coagulopathy.
  * Emergency cesarean section.
  * Failed or unsatisfactory intrathecal block.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 204 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
severity of pruritus that occurs after intrathecal morphine in parturient undergoing elective cesarean section (CS) by pruritus Grading system. | 24 hours
  the pruritus grading score (PGS) score (Firas et al, 2012) for each patient which is based on: distribution, frequency, severity of itch, and quality of sleep
  Each patient's itch grade is calculated as the sum of the individual scores:
  Mild grade: if the total score is between 0 and 5. Moderate grade: if the total score is between 6 and 11. Severe grade: if the total score is between 12 and 19.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kumar K, Singh SI. Neuraxial opioid-induced pruritus: An update. J Anaesthesiol Clin Pharmacol. 2013 Jul;29(3):303-7. doi: 10.4103/0970-9185.117045. PMID 24106351
- [Result] Singh PM, Sultan P, O'Carroll J, Blake L, Carvalho B, Singh NP, Monks DT. Pharmacological agents for prevention of pruritus in women undergoing Caesarean delivery with neuraxial morphine: a systematic review and Bayesian network meta-analysis. Br J Anaesth. 2023 Sep;131(3):556-571. doi: 10.1016/j.bja.2023.05.028. Epub 2023 Jul 14. PMID 37455197
- [Result] Kampo S, Afful AP, Mohammed S, Ntim M, Buunaaim ADB, Anabah TW. Sub-hypnotic dose of propofol as antiemetic prophylaxis attenuates intrathecal morphine-induced postoperative nausea and vomiting, and pruritus in parturient undergoing cesarean section - a randomized control trial. BMC Anesthesiol. 2019 Sep 14;19(1):177. doi: 10.1186/s12871-019-0847-y. PMID 31521119